CLINICAL TRIAL: NCT01742494
Title: Peroral Endoscopic Myotomy for Esophageal Achalasia: Randomized Comparison of Water-Jet Assisted Versus Conventional Dissection Technique
Brief Title: Comparison Study of Conventional POEM and Hybrid POEM for Esophageal Achalasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hybrid POEM
Record Dates: First submitted 2012-11-20; First posted 2012-12-05 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Esophageal Achalasia
Keywords: Esophageal Achalasia,; Peroral endoscopic myotomy,; Water-jet assisted
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Water-jet POEM (Active Comparator): POEM were performed by the use of Erbe Hybrid knife (WJ group)
  Interventions: Procedure: Water-jet POEM
- Conventional POEM (Active Comparator): POEM were performed by the conventional technique using injection and triangle tip knife (C group).
  Interventions: Procedure: Conventional POEM

INTERVENTIONS:
Procedure: Water-jet POEM — Water-jet assisted POEM procedure was performed
  Arms: Water-jet POEM
Procedure: Conventional POEM — POEM were performed by the use of conventional technique using injection and triangle tip knife.
  Arms: Conventional POEM

SUMMARY:
Peroral endoscopic myotomy (POEM) has recently been introduced as promising alternative to laparoscopic Heller myotomy for patients with idiopathic achalasia. Several technical modifications have been proposed but have not yet been tested in randomized trials.

DETAILED DESCRIPTION:
Objective: To evaluate efficacy and safety of water-jet assisted POEM (WJ) versus the conventional technique (C).

Interventions: Patients with achalasia diagnosed by symptoms, endoscopy and barium swallow eligible for POEM were randomized to either the use of Erbe Hybrid knife (WJ group) or the conventional technique using injection and triangle tip knife interchangeably (C group).

Main outcome measurements: Procedure time in both groups; secondary outcomes were clinical efficacy and safety (bleeding complications, pneumothorax or pleural effusion requiring intervention)

ELIGIBILITY:
Inclusion Criteria:

* With an Eckardt symptom score ≥ 4
* The diagnosis of achalasia was made on the basis of the absence of peristalsis and on impaired relaxation of the LES on established methods (barium swallow, manometry, esophagogastroduodenoscopy)
* Informed patient consent was obtained

Exclusion Criteria:

* Severe cardiopulmonary disease or other serious disease leading to unacceptable surgical risk
* Pseudoachalasia
* Megaesophagus (diameter of > 7 cm)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Procedure time in both groups | during POEM procedure

SECONDARY OUTCOMES:
clinical efficacy and safety | during hospital stay and up to 1 year
  bleeding complications, pneumothorax or pleural effusion requiring intervention

OTHER OUTCOMES:
Therapeutic success | Every 3 months after innitial intervention via telephone questionnaires during follow-up up to 1 year
  a reduction in the Eckardt score to ≤3

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Hong Zhou, M.D., PhD, Study Director — Fudan University
Locations (1):
- Endoscopy Center and Endoscopy Research Institute, Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Cai MY, Zhou PH, Yao LQ, Xu MD, Zhong YS, Li QL, Chen WF, Hu JW, Cui Z, Zhu BQ. Peroral endoscopic myotomy for idiopathic achalasia: randomized comparison of water-jet assisted versus conventional dissection technique. Surg Endosc. 2014 Apr;28(4):1158-65. doi: 10.1007/s00464-013-3300-1. PMID 24232052